CLINICAL TRIAL: NCT00092391
Title: A Study of M-M-R(TM) II at Mumps Expiry Potency in Healthy Children 12 to 18 Months of Age
Brief Title: A Study of An Approved Vaccine at Mumps Expiry Potency in Healthy Children 12 to 18 Months of Age (V205C-007)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: V205C-007; 2004_073
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — Rubella Vaccine; Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Control Group (Active Comparator): M-M-R(TM) II at current release potency
  Interventions: Biological: Comparator: M-M-R(TM) II, measles, mumps, and rubella virus vaccine live; Biological: Comparator: VARIVAX(TM) Varicella Virus Vaccine Live (Oka-Merck)
- Mumps Expiry Group 1 (Experimental): M-M-R(TM) II at intermediate expiry potency
  Interventions: Biological: Comparator: M-M-R(TM) II, measles, mumps, and rubella virus vaccine live; Biological: Comparator: VARIVAX(TM) Varicella Virus Vaccine Live (Oka-Merck)
- Mumps Expiry Group 2 (Experimental): M-M-R(TM) II at expiry potency
  Interventions: Biological: Comparator: M-M-R(TM) II, measles, mumps, and rubella virus vaccine live; Biological: Comparator: VARIVAX(TM) Varicella Virus Vaccine Live (Oka-Merck)

INTERVENTIONS:
Biological: Comparator: M-M-R(TM) II, measles, mumps, and rubella virus vaccine live — 0.5 mL subcutaneous injection of one of three sub-lots on Day 0
Biological: Comparator: VARIVAX(TM) Varicella Virus Vaccine Live (Oka-Merck) — 0.5 mL subcutaneous injection on Day 0

SUMMARY:
The purpose of this study is to determine the mumps virus strength at the end of shelf-life (expiration date) of an approved vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 12 to 18 months of age

Exclusion Criteria:

* History or prior exposure to measles, mumps, rubella or varicella
* History of anaphylactoid reactions or hypersensitivity to any component of the vaccine, including gelatin and neomycin

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1997 (Actual)
Dates: Start 1999-02; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Neutralizing antibodies to mumps at 6 weeks postvaccination | 6 weeks postvaccination

SECONDARY OUTCOMES:
Geometric mean titers to mumps by ELISA at 6 weeks and at 1 year postvaccination | 6 weeks and 1 year postvaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC